CLINICAL TRIAL: NCT02638064
Title: Treatment of Pilonidal Sinus Disease Using Surgiflo as a Sealant: A New Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mansourau25
Record Dates: First submitted 2015-10-29; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Pilonidal Sinus Disorder
MeSH Terms: interventions — Surgiflo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgiflo injection (Experimental): Injection of surgiflo in the pilonidal sinus cavity after curettage of its content
  Interventions: Procedure: Surgiflo injection

INTERVENTIONS:
Procedure: Surgiflo injection — Curettage of sinus cavity then injection of surgiflo material

SUMMARY:
Assessment of surgiflo injection for treating pilonidal sinus disease

DETAILED DESCRIPTION:
Evaluation of injection of Surgiflo as a sealent in treatment of pilonidal sinus, evaluation includes recurrence, infection, complications and patient satisfaction over 2 years of follow up

ELIGIBILITY:
Inclusion Criteria:

Patients included in the study had simple midline PS with single or multiple tracts and no lateral extensions. Recurrent cases of PS after previous surgery were also included in the study

Exclusion Criteria:

We excluded from the study patients with severe scarring at the natal cleft due to previous surgery or infection and patients with signs of an acute abscess.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of the condition | 2 years
  number of patients presenting with recurrent pilonidal sinus

SECONDARY OUTCOMES:
Complications of the procedure | 2 years
  number of patients presenting with complications after injection of surgiflo

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Elbanna, M.D, Principal Investigator — private basis
Locations (1):
- Hosam Elbanna, Al Mansurah, Dakahlia Governorate, Egypt